CLINICAL TRIAL: NCT06278922
Title: Evaluating Signs of Safety: A Deaf-Accessible Therapy Toolkit for AUD and Trauma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Melissa L. Anderson, Associate Professor of Psychiatry, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00001149; R01AA031010 (NIH)
Record Dates: First submitted 2024-02-17; First posted 2024-02-26 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: PTSD; Alcohol; Use, Problem
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Alcoholism | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The PI will be masked to study condition. All outcome data will be collected via online self-report surveys.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Seeking Safety + Signs of Safety toolkit (Experimental): Experimental participants will be offered 12 one-hour, weekly individual therapy sessions of Seeking Safety delivered with the Signs of Safety toolkit. Sessions will occur virtually via National Deaf Therapy's (NDT) secure HIPAA-compliant video chat platform. Length of treatment is limited to six months; number of completed sessions will be tracked as a measure of participant adherence.
  Interventions: Behavioral: Seeking Safety + Signs of Safety toolkit
- Treatment as usual (Active Comparator): Participants assigned to the active comparison condition will receive therapy as usual - i.e., general, open-ended, non-manualized supportive counseling provided by an NDT therapist. In the absence of any evidence-based therapies available for Deaf clients, this unstructured therapy approach is the current standard of care in the field of Deaf mental health. All NDT therapists are Deaf, fluent in ASL, and specialize in issues common to Deaf individuals seeking mental health care. Like the experimental condition, participants will receive 12 one-hour, weekly individual therapy sessions via NDT's secure virtual therapy platform. Length of treatment is limited to six months; number of completed sessions will be tracked as a measure of participant adherence.
  Interventions: Behavioral: Treatment as usual
- No treatment (No Intervention): Participants in states with no NDT therapists and who prefer to be placed on NDT's waitlist instead of being referred outside of NDT for therapy will be automatically assigned to the no-treatment control condition. At the time of this submission, there are approximately 200 individuals on the NDT waitlist; individuals remain on the waitlist until a licensed therapist from their state joins the NDT team. Participants in the control condition will be prompted to complete assessments at baseline, week 6, week 12 (to approximate immediate post-treatment), week 25 (to approximate three-month follow-up), and week 38 (to approximate six-month follow-up). Such repeated assessment in the control arm will allow us to quantify and control for participants' natural change over time and any potential assessment reactivity.

INTERVENTIONS:
Behavioral: Seeking Safety + Signs of Safety toolkit — Signs of Safety is a Deaf-accessible toolkit to be used with the Seeking Safety treatment protocol. Seeking Safety is a manualized, non-exposure-based, cognitive behavioral therapy for trauma and addiction.
  Arms: Seeking Safety + Signs of Safety toolkit
Behavioral: Treatment as usual — NDT therapists come from a wide variety of training backgrounds, but each works with their clients to build on their existing strengths and provide support as clients develop new strategies and behaviors for overcoming adversity.
  Arms: Treatment as usual

SUMMARY:
The U.S. Deaf community - a group of more than one million Americans who communicate using American Sign Language (ASL) - experiences nearly triple the rate of lifetime problem drinking and twice the rate of trauma exposure compared to the general population. Although there are several treatments for alcohol use disorder (AUD) and posttraumatic stress disorder (PTSD) in hearing populations, none have been developed for or tested with Deaf clients. To address these barriers, the study team developed Signs of Safety, a Deaf-accessible therapy toolkit for treating AUD and PTSD. Their aims are to conduct a nationwide, virtual clinical trial to compare (1) Signs of Safety with (2) treatment as usual and (3) a no treatment control, to collect data on clinical outcomes, and to explore potential mediators and moderators of outcome.

DETAILED DESCRIPTION:
In partnership with Deaf-owned agency National Deaf Therapy, the study team will conduct the first-ever full-scale psychotherapy trial conducted in the Deaf community - "Evaluating Signs of Safety: A Deaf-Accessible Therapy Toolkit for AUD and Trauma." The U.S. Deaf community - more than one million Americans who communicate using American Sign Language (ASL) - experiences nearly triple the rate of lifetime problem drinking compared to the general population (33.0% vs. 12.3%) and twice the rate of trauma exposure. Among Deaf people in treatment for alcohol use disorder (AUD), 74% report lifetime physical, emotional, or sexual abuse and 44% report past-year abuse. Comorbid AUD/PTSD impairs multiple domains of functioning, especially for Deaf individuals, who show poorer functional outcomes than hearing individuals in socialization, employment, and physical health.

Hearing individuals have access to several validated treatments for comorbid AUD/PTSD; yet there are no evidence-based treatments to treat any behavioral health condition with Deaf clients. Available treatments fail to meet Deaf clients' unique language access needs. Deaf people's median English literacy level falls at the fourth grade and health-related vocabulary among Deaf sign language users parallels non-English-speaking U.S. immigrants. Available treatment resources, therefore, require plain text revisions, filmed ASL translations, or education through storytelling to better match Deaf clients' language needs.

Leveraging extensive community engagement to address these barriers, the Principal Investigator's team of Deaf and hearing researchers, clinicians, filmmakers, actors, artists, and Deaf people with AUD/PTSD developed and pilot tested Signs of Safety, a Deaf-accessible toolkit to be used with the Seeking Safety treatment protocol. Seeking Safety is a manualized, non-exposure-based, cognitive behavioral therapy for trauma and addiction. Among evidence-based treatments for AUD/PTSD, Seeking Safety is the optimal choice for Deaf clients - its focus on psychoeducation and simple coping skills is an ideal match for Deaf people's language and literacy disparities, which prohibit the use of narrative, verbal problem-solving, and cognitive processing strategies that other AUD/PTSD therapies require. Yet, Seeking Safety's client materials rely on written English and are, therefore, not well understood by Deaf clients. As such, the Signs of Safety toolkit provides a supplemental therapist guide and population-specific client materials (e.g., visual handouts, filmed ASL teaching stories).

Preliminary data from the Signs of Safety single-arm pilot and randomized feasibility pilot showed reductions in alcohol use frequency and PTSD severity from baseline to follow-up on the Reliable Change Index. The delivery of the experimental intervention was deemed feasible by study therapists and was well-received by participants, especially when moved to a virtual platform. In response to the COVID-19 pandemic, the study team overhauled in-person study methods to implement a virtual clinical trial - an acceleration of the inevitable development needed to scale Signs of Safety to a national level. This adaptation also established a crucial collaboration with National Deaf Therapy (NDT), by far the nation's largest provider of Deaf mental health services, currently serving clients across 21 states. This collaboration, paired with comprehensive feasibility data the study team collected by testing a variety of virtual methods, serves as the foundation of the study team's proposed aims.

The study team will conduct a nationwide, full-scale, virtual clinical trial of Signs of Safety. Leveraging the existing infrastructure and robust referral network of NDT, the study team will enroll 144 Deaf adults with past-month PTSD and problem drinking. Primary clinical outcomes at immediate post-treatment are change from baseline percent binge drinking days per month (Alcohol Timeline Followback) and change from baseline past 30-day PTSD severity (PTSD Checklist for DSM-5). Assessment will occur at baseline, mid-treatment, immediate post-treatment, three-month post-treatment follow-up, and six-month post-treatment follow-up. Participants residing in states served by NDT (n = 96) will be randomized to receive either (1) a 12-session protocol of Seeking Safety + Signs of Safety, or (2) 12 sessions of therapy as usual (TAU; general, open-ended, non-manualized supportive counseling provided by an NDT therapist). The study team will enroll an additional 48 Deaf adults into a contemporaneous no-treatment control arm. These individuals will be recruited from the existing NDT waitlist, comprised of Deaf individuals residing in the states not yet served by NDT but voluntarily awaiting NDT services. Additionally, the study team will analyze potential moderators and mediators that lead to positive outcome. Identified from the literatures on Seeking Safety, alcohol treatment research, and Deaf mental health research, mechanisms of change are coping self-efficacy, self-compassion, motivation for treatment, and access to health information.

They study team's proposed aims build upon eight years of empirical work, moving the program of research from Stage IB (two-arm feasibility and pilot testing) to Stage II/III (real world efficacy). This clinical trial will potentially validate the first-ever evidence-based therapy for Deaf people, as well as provide future behavioral health researchers with a vital roadmap for conducting community-engaged clinical trials with Deaf people.

ELIGIBILITY:
Inclusion Criteria:

* Self-identification as Deaf or hard-of-hearing
* Proficiency in American Sign Language (ASL)
* Age 18 years or older
* Access to videoconferencing technology for informed consent and, if applicable, study therapy sessions
* Access to online survey technology for study assessments
* "Problematic alcohol consumption, drinking behaviors, and alcohol-related problems" on the AUD Identification Test (AUDIT), a 10-item screening measure developed by the World Health Organization that demonstrates good sensitivity and specificity in many populations (past-month referent time period; score ≥ 8 for men or ≥ 6 for women)
* "Subthreshold or full PTSD," on the PTSD Checklist for DSM-5 (PCL-5), a 20-item measure of PTSD symptoms reliably used to monitor symptom change (past-month referent time period; "subthreshold" = meets at least two DSM-5 diagnostic categories (B, C, D, and/or E) at moderate or high severity)

Exclusion Criteria:

* Participation in concurrent formal psychotherapy (Note: Participants in all study conditions will be asked to refrain from concurrent formal psychotherapy. Participants who engage in formal psychotherapy outside of the research will be removed from the study at the point of treatment initiation. Outside treatment engagement will be queried at each assessment timepoint. If endorsed, the participant will be removed from the study at that timepoint, but data collected prior to treatment initiation will remain in the dataset. Aligning with the Seeking Safety model, Alcoholics Anonymous/Narcotics Anonymous/Dual Recovery Anonymous attendance will be encouraged; attendance will be tracked as a potential outcome mediator.)
* Members of the following special populations: Adults unable to consent; Individuals younger than 18 years; Prisoners; Pregnant women (Note: The investigators will not knowingly include pregnant women as participants; however, the investigators will not assess participants' pregnancy status.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2024-12-23 (Actual); Primary Completion 2028-11-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Percent Binge Drinking Days Per Month at Immediate Post-Treatment as Measured by the Alcohol Timeline Followback | Change from baseline to immediate post-treatment at 12 weeks
  Change from baseline percent binge drinking days per month (i.e., days with 5+ drinks for men, 4+ for women) at immediate post-treatment or 12 weeks as assessed by the Alcohol Timeline Followback
Change from Baseline Past 30-day PTSD Severity to Immediate Post-Treatment as Measured by the PCL-5 | Change from baseline to immediate post-treatment at 12 weeks
  Total Score on the PCL-5 divided by 20 items. Minimum score = 0; Maximum score = 4. Higher values represent more severe symptoms of PTSD.

SECONDARY OUTCOMES:
Change from Baseline Percent Drinking Days Per Month at Immediate Post-Treatment as Measured by the Alcohol Timeline Followback | Change from baseline to immediate post-treatment at 12 weeks
  Change from baseline percent drinking days per month (i.e., days with 1+ drink) at immediate post-treatment or 12 weeks as assessed by the Alcohol Timeline Followback
Change from Baseline Percent Drinking Days Per Month at Three-month Follow-up as Measured by the Alcohol Timeline Followback | Change from baseline to three-month follow-up at 25 weeks
  Change from baseline percent drinking days per month (i.e., days with 1+ drink) at three-month follow-up or 25 weeks as assessed by the Alcohol Timeline Followback
Change from Baseline Percent Drinking Days Per Month at Six-month Follow-up as Measured by the Alcohol Timeline Followback | Change from baseline to six-month follow-up at 38 weeks
  Change from baseline percent drinking days per month (i.e., days with 1+ drink) at six-month follow-up or 38 weeks as assessed by the Alcohol Timeline Followback
Change from Baseline Percent Binge Drinking Days Per Month at Three-month Follow-up as Measured by the Alcohol Timeline Followback | Change from baseline to three-month follow-up at 25 weeks
  Change from baseline percent binge drinking days per month (i.e., days with 5+ drinks for men, 4+ for women) at three-month follow-up or 25 weeks as assessed by the Alcohol Timeline Followback
Change from Baseline Percent Binge Drinking Days Per Month at Six-month Follow-up as Measured by the Alcohol Timeline Followback | Change from baseline to six-month follow-up at 38 weeks
  Change from baseline percent binge drinking days per month (i.e., days with 5+ drinks for men, 4+ for women) at six-month follow-up or 38 weeks as assessed by the Alcohol Timeline Followback
Change from Baseline Number of Drinks Per Month at Immediate Post-Treatment as Measured by the Alcohol Timeline Followback | Change from baseline to immediate post-treatment at 12 weeks
  Change from baseline number of drinks per month at immediate post-treatment or 12 weeks as assessed by the Alcohol Timeline Followback
Change from Baseline Number of Drinks Per Month at Three-month Follow-up as Measured by the Alcohol Timeline Followback | Change from baseline to three-month follow-up at 25 weeks
  Change from baseline number of drinks per month at three-month follow-up or 25 weeks as assessed by the Alcohol Timeline Followback
Change from Baseline Number of Drinks Per Month at Six-month Follow-up as Measured by the Alcohol Timeline Followback | Change from baseline to six-month follow-up at 38 weeks
  Change from baseline number of drinks per month at six-month follow-up or 38 weeks as assessed by the Alcohol Timeline Followback
Change from Baseline Past 30-day PTSD Severity to Three-month Follow-up as Measured by the PCL-5 | Change from baseline to three-month follow-up at 25 weeks
  Total Score on the PCL-5 divided by 20 items. Minimum score = 0; Maximum score = 4. Higher values represent more severe symptoms of PTSD.
Change from Baseline Past 30-day PTSD Severity to Six-month Follow-up as Measured by the PCL-5 | Change from baseline to six-month follow-up at 38 weeks
  Total Score on the PCL-5 divided by 20 items. Minimum score = 0; Maximum score = 4. Higher values represent more severe symptoms of PTSD.
Change from Baseline Diagnostic and Statistical Manual (DSM)-5 diagnostic criteria for Alcohol Use Disorder to Immediate Post-Treatment as measured by the DSM-5 AUD Assessment Tool | Change from baseline to immediate post-treatment at 12 weeks
  Total Score on the DSM-5 AUD Assessment Tool. Minimum score = 0; Maximum score = 13. Higher values represent more severe symptoms of AUD.
Change from Baseline Percent Days of Drug Use Per Month at Immediate Post-Treatment as Measured by the Timeline Followback - Drugs, Cigarettes, and Marijuana | Change from baseline to immediate post-treatment at 12 weeks
  Change from baseline percent drug use days per month (i.e., days with 1+ drug) at immediate post-treatment or 12 weeks as assessed by the Timeline Followback - Drugs, Cigarettes, and Marijuana
Change from Baseline Number of Instances of Drug Use Per Month at Immediate Post-Treatment as Measured by the Timeline Followback - Drugs, Cigarettes, and Marijuana | Change from baseline to immediate post-treatment at 12 weeks
  Change from baseline number of instances of drug use per month at immediate post-treatment or 12 weeks as assessed by the Timeline Followback - Drugs, Cigarettes, and Marijuana
Change from Baseline Percent Days of Marijuana Use Per Month at Immediate Post-Treatment as Measured by the Timeline Followback - Drugs, Cigarettes, and Marijuana | Change from baseline to immediate post-treatment at 12 weeks
  Change from baseline percent marijuana use days per month (i.e., days with 1+ instance of marijuana use) at immediate post-treatment or 12 weeks as assessed by the Timeline Followback - Drugs, Cigarettes, and Marijuana
Change from Baseline Number of Instances of Marijuana Use Per Month at Immediate Post-Treatment as Measured by the Timeline Followback - Drugs, Cigarettes, and Marijuana | Change from baseline to immediate post-treatment at 12 weeks
  Change from baseline number of instances of marijuana use days per month at immediate post-treatment or 12 weeks as assessed by the Timeline Followback - Drugs, Cigarettes, and Marijuana
Change from Baseline Percent Days of Tobacco Use Per Month at Immediate Post-Treatment as Measured by the Timeline Followback - Drugs, Cigarettes, and Marijuana | Change from baseline to immediate post-treatment at 12 weeks
  Change from baseline percent tobacco use days per month (i.e., days with 1+ instance of tobacco use) at immediate post-treatment or 12 weeks as assessed by the Timeline Followback - Drugs, Cigarettes, and Marijuana
Change from Baseline Number of Instances of Tobacco Use Per Month at Immediate Post-Treatment as Measured by the Timeline Followback - Drugs, Cigarettes, and Marijuana | Change from baseline to immediate post-treatment at 12 weeks
  Change from baseline number of instances of tobacco use days per month at immediate post-treatment or 12 weeks as assessed by the Timeline Followback - Drugs, Cigarettes, and Marijuana
Change from Baseline Substance-related Problems at Immediate Post-Treatment as Measured by the Short Inventory of Problems Revised (SIPS-R) | Change from baseline to immediate post-treatment at 12 weeks
  Total Score on the SIPS-R. Minimum score = 0; Maximum score = 51. Higher values represent more severe substance-related problems.
Change from Baseline Alcohol Craving at Immediate Post-Treatment as Measured by the Brief Addiction Monitor - Revised (BAM-R) | Change from baseline to immediate post-treatment at 12 weeks
  One-item measure of craving from the BAM-R, scored from 0 ("not at all") to 4 ("extremely"). Higher values represent more severe levels of craving.
Change from Baseline Drug Craving at Immediate Post-Treatment as Measured by the Brief Addiction Monitor - Revised (BAM-R) | Change from baseline to immediate post-treatment at 12 weeks
  One-item measure of craving from the BAM-R, scored from 0 ("not at all") to 4 ("extremely"). Higher values represent more severe levels of craving.
Change from Baseline Marijuana Craving at Immediate Post-Treatment as Measured by the Brief Addiction Monitor - Revised (BAM-R) | Change from baseline to immediate post-treatment at 12 weeks
  One-item measure of craving from the BAM-R, scored from 0 ("not at all") to 4 ("extremely"). Higher values represent more severe levels of craving.
Change from Baseline Tobacco Craving at Immediate Post-Treatment as Measured by the Brief Addiction Monitor - Revised (BAM-R) | Change from baseline to immediate post-treatment at 12 weeks
  One-item measure of craving from the BAM-R, scored from 0 ("not at all") to 4 ("extremely"). Higher values represent more severe levels of craving.
Change from Baseline Psychosocial Functioning at Immediate Post-Treatment as Measured by the Outcome Questionnaire (OQ-30.2) for Adults | Change from baseline to immediate post-treatment at 12 weeks
  Total Score on the OQ-30.2. Minimum score = 0; Maximum score = 120; Clinical cutoff = greater than or equal to 44. Higher values represent higher levels of psychosocial distress related to experiencing a high number of symptoms, interpersonal difficulties, and/or decreased satisfaction and quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Massachusetts Medical School, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators will submit and share data with the NIAAA Data Archive, a data repository housed within the National Institute on Mental Health (NIMH) Data Archive (NDA), per the requirements set forth in NOT-AA-23-002 (grants.nih.gov/grants/guide/notice-files/NOT-AA-23-002.html). All data will be de-identified before submission to the data archive.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The investigators will submit data on or before the NDA submission due dates (April 1 and October 1 each year) in accordance with the applicable Data Sharing Terms and Conditions of award.
Access Criteria: Can be accessed via the NIAAA Data Archive (NIAAADA)
URL: https://nda.nih.gov/niaaa

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-02-16): https://cdn.clinicaltrials.gov/large-docs/22/NCT06278922/Prot_SAP_000.pdf
  • Informed Consent Form (2023-08-21): https://cdn.clinicaltrials.gov/large-docs/22/NCT06278922/ICF_001.pdf